CLINICAL TRIAL: NCT03357042
Title: A Multi-modal Evaluation of a Physical Intervention Approach to Treating Post-Concussive Symptoms
Brief Title: Evaluation of a Physical Intervention for Persistent Post-Concussive Symptoms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: researchers did not find participants to meet the inclusion and exclusion criteria for the testing protocols
Sponsor: Lakehead University (Other)
Collaborators: Northern Ontario School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP-506-07112017
Record Dates: First submitted 2017-11-09; First posted 2017-11-29 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2019-08

CONDITIONS: Persistent Post-Concussive Syndrome
MeSH Terms: interventions — Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: Three group: Aerobic retraining intervention, standard of care intervention, healthy control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Persistent post-concussive symptoms (Experimental): Participants who report post-concussive symptoms. 20 participants will receive the aerobic exercise and balance training intervention, 20 participants will receive standard of care treatment for concussions.
  Interventions: Other: Aerobic exercise and balance retraining; Other: Standard of care
- Healthy control (Active Comparator): Persons without post-concussive symptoms. No intervention.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Aerobic exercise and balance retraining — Aerobic and balance exercises that gradually progress in intensity over the course of 8 weeks.
  Arms: Persistent post-concussive symptoms
Other: Standard of care — Normal concussion treatment; physical and cognitive rest

SUMMARY:
A concussion occurs when a person receives an impact to the head. The most common persistent symptoms that generate from a concussion are headaches, depression, lack of balance and dizziness. One recommendation to alleviate persistent symptoms of concussion is rest. Research findings indicate that the benefit of rest is inconclusive to help individuals suffering from a concussion return to activities of daily living. One treatment approach in reducing concussion symptoms is physical exercise therapy. Research findings, however, are limited to treatments being administered before the symptoms are considered persistent. Based on this rationale, the aim of this study is to examine the effect of a physical therapy intervention in minimizing persistent symptoms of concussion using measures of cognition and brain function, mental and physical health, and driving performance. If successful, this physical therapy intervention may help treat persistent concussion symptoms, improving the quality of life and ability for individuals to function normally in their daily lives, and resulting in savings to the healthcare system

DETAILED DESCRIPTION:
Recruitment will include the use of posters, social media, and word of mouth. Posters designed to recruit healthy individuals free of a concussion will be displayed around Lakehead University, as well as various public spaces in Thunder Bay. Separate posters (attached) will also be used to recruit persons who have sustained a concussion in the previous two weeks to six months and are still experiencing symptoms (Persistent Post-concussive symptoms; PCS). These posters will be displayed at Fairway Physiotherapy and healthcare clinics around Thunder Bay. All posters will be shared on Lakehead University School of Kinesiology social media pages.

Prior to participating in the study, all participants will have a medical examination with Dr. Wark at least two weeks following the initial injury. If the potential participant expresses interest in the study, his/her information will be passed along to a member of the research team. A member of the research team will contact the potential participant to schedule pre intervention assessments based on the participant's, research team, and lab availability. Participants will also be provided with a copy of the information letter at this time. Any medical screening tools will be kept by Dr. Wark as part of the patient's medical records, regardless of eligibility for the study. Any information taken from these records will be recorded using a data abstraction form.

Healthy and PCS participants will be scheduled for pre intervention physical, cognitive, neuroimaging, biomarker, and driving behaviour assessments at Lakehead University. All pre intervention assessments will be completed over the course of one week. At the first session, a member of the research team will complete the informed consent process; participants will be provided with a verbal overview of the study and the information letter. Following the informed consent process, healthy participants will complete the short form International Physical Activity Questionnaire.

Following the informed consent process, PCS participants will be provided with Garmin VivoSmart heart rate (HR) unit to monitor aerobic activity outside of the study (accelerometer, heart rate monitor, and step counter capabilities). Participants will be required to wear the Garmin units as often as possible for the duration of the study. Depending on scheduling, participant's will then complete one of the baseline assessments.

Baseline Assessments

Physical and Cognitive Assessment:

Participants will complete the Immediate Post-concussion Assessment and Cognitive Testing (ImPACT) at the School of Kinesiology, Sanders building, Lakehead University. The ImPACT will be used as a question and answered based, standard measure of cognitive abilities including: attention, working memory, processing speed, and reaction time. Following completion of the ImPACT battery, participants will be asked to stand in a variety of static positions including: narrow based double leg stance, single leg stance, and tandem stance with one foot behind the other. Participants will perform each stance position with his/her eyes open and closed and on a firm and soft surface using the Balance Error Scoring System (BESS) protocol. Each stance will be performed over an Advanced Medical Technologies Incorporated (AMTI) force platform. The session should last approximately one hour.

Biomarker Assessment:

Brain-derived neurotropic factor (BDNF) will be assessed using a morning saliva sample. Participants will be asked to refrain from brushing his/her teeth, smoking, and consuming food or drink within two hours of the sample collection. Participants will also be asked to avoid alcohol consumption 12 hours prior to sampling. At a mutually agreed upon date and time, the participant will meet a member of the research team at the School of Kinesiology, Sanders building, Lakehead University. Before beginning saliva collection, the member of the research team will verbally restate the participant's rights and confirm that he/she is still willing to participate in the study. Saliva will then be collected from participants in room SB-1025 (biohazard containment level 1) via the passive drool method into a tube, which will then be transported to Dr. Lees lab for processing.

Neuroimaging:

Neural processing will be assessed by using continuously recorded electroencephalography (EEG) during the performance of computer based tasks commonly used in experimental psychology for assessing divided attention and inhibitory control. Participants will be seated at a desk and fitted with an EEG cap and 32 channels will be prepared with gel. Once all recording sites are ready for recording the participant will be familiarized with the task procedures and equipment. At the desk he/she is seated at, he/she will view a monitor and be provided with a response pad. Participants will complete the Oddball paradigm and Flanker task. Completion of the session should require two hours.

Tasks:

ODDBALL paradigm:

The Oddball paradigm is a commonly used task to test attention by requiring participants to make a specific response to rare target stimuli amongst more repetitive, distractor stimuli (Squires, Squires, & Hillyard, 1975). In this visual version, participants will be provided an instruction at the outset of a block that indicates what the target stimulus for that block will be. During each trial, a stimulus (shape/letter) will be displayed for 200 milliseconds (ms). Participants will be instructed to respond to each stimulus as quickly and accurately as possible with a button press of one of two buttons; a button to denote distractor stimuli, and a button to indicate target stimuli. The interstimulus interval will be variable (1400-1600 ms) to reduce anticipation. Participants will complete 400 trials separated into 5 blocks with an option for rests between each block.

FLANKER task:

The Flanker task is commonly used to test the ability to attend to central relevant information (the direction of an arrow) while disregarding irrelevant distracting stimuli (pairs of flanking arrows presented on either side of the central arrow). To identify the direction of the central arrow, participants will press a left or right button to indicate the direction of the central arrow. Data will be separated into time frames containing the components of interest (the N200 and P300). The session is concluded after completion of the oddball and flanker tests twice.

Behaviour Measure (Driving Simulator):

The performance of participants in a driving simulator will be assessed by measuring his/her reaction time and counting the number of passes and failures when anticipating potentially dangerous traffic situations. Reaction time will also be measured during dual-tasking activities.

Participants will perform a 10 minute orientation drive to familiarized his/herself with the control and feel of the driving simulator. During the orientation drive, he/she will be exposed to examples of the dual tasking activities so that he/she will know how to successfully respond to the prompts. Once a participant feels comfortable with the simulator, the 20 minute simulation and data collection will begin. The simulation will be based on the Thunder Bay road system with traffic and pedestrians present. Weather will be clear and visibility will not be reduced. Reaction times will be measured during predetermined scenarios and will be recorded from the moment stimulus occurs to the moment the brake is depressed or evasive maneuver performed. Participants will be exposed to several scenarios. These scenarios include: Vehicle incursion at intersection, pedestrian incursion from side of the road, sudden braking by a vehicle in front of participant, pedestrian incursion in school zone, braking by a vehicle in front of participant, and animal incursion (attached)

During dual task events, red triangles will be displayed over either of the side mirrors. These triangles will be deactivated by the press of a button on either side of the steering column, accounting for the dual tasking component of the reaction time scenarios The research team member will have water on hand, if required by the participant. When he/she feels ready to proceed, the simulation will be resumed from the point of the original pause. If a participant feels that he/she is unable to continue, the simulation will be stopped and data collection terminated.

Randomization Prior to the implementation of the interventions, PCS participants will be randomly assigned to either an AET or standard of care (SC) intervention. Using minimization software, each intervention group will be balanced by sex and age. Healthy participants will serve as the control group (HC) and will receive no treatment. Once participants in the SC group have completed the study, the AET will be offered, although it will not be included in the data analysis. All participant information/group assignment will be coded to maintain confidentiality.

Aerobic and Balance Retraining Program:

After completing baseline assessments, PCS participants assigned to the aerobic and balance retraining (AET) intervention will complete an eight week supervised AET program. The program will consist of three sessions per week, approximately 40-60 minutes each. Each session will be performed under the supervision of a trainer that has the Canadian Society for Exercise Physiology (CSEP-CPT) certification.

The aerobic component of the session will be performed on a cycle ergometer. Participants will begin with a five minute warmup at a self selected speed, which will be used to bring the participant's heart rate to the desired intensity. Intensity for each session will start at 20% of heart rate reserve (HRR), and increase linearly by 10% for the first four weeks; at week four, participants will be cycling at an intensity of 50%. Weeks five and six will be performed at 55% of HRR, week seven will be performed at 60% of HRR, and week eight will be performed at 65% of HRR. Duration will follow a similar pattern for weeks one to four, beginning at 20 minutes and increasing in five minutes/week increments. At week five, duration will be reduced to 25 minutes, and then increase to 30 minutes for weeks six to eight.

Following completion of the aerobic portion of the session, participants will rest for five minutes before beginning the balance component of the session. Participants will perform three balance exercises (in order) each session: narrow based double leg stance, single leg stance, and tandem stance. Difficulty of these exercises will be progressively increased by modifying the duration, surface, and whether the participant's eyes are open or closed. For weeks one and two participants will perform the exercises with his/her eyes open; participants will perform each exercise for 15 seconds on a firm service in week one, and on a low density foam block in week two. In weeks three and four, participants will perform the exercises with his/her eyes closed; exercises in week three will be performed on a firm surface, while week four will be performed on a low density foam block. Duration will be increased to twenty seconds per exercise for weeks three and four. Weeks four to eight will follow the same eyes open/closed and surface progression as weeks one to four; eyes open for weeks five and six, eyes closed for weeks seven and eight. Exercises will be performed on a firm surface in weeks five and seven, and on a low density foam block in weeks six and eight. Participants will perform each exercise for 35 seconds in weeks five and six, and 40 seconds in weeks seven and eight. Following the completion of the aerobic and balance components of the session, participants will complete a cool down consisting of a series of static stretches. Each session will conclude after the completion of the cooldown.

After completion of 24 sessions (eight weeks x three-one hour sessions per week), participants will repeat the procedures for the previously described baseline assessments. Similarly, HC and SC participants will complete the baseline assessments again after eight weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged 18-50 years.
2. Reports at least one PCS symptom that is mild in severity.
3. It has been two weeks since date of injury.

Exclusion Criteria:

1. Has been previously diagnosed with a psychological/neurological disorder
2. Has been previously diagnosed with a substance abuse disorder/impairment,
3. Is currently seeking therapy/counseling
4. Does not have valid driver's license and 12 months of driving experience.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Star Excursion Balance Test (SEBT) | 8 weeks
  Measure of balance. Score is based on normalized percentage of maximum reach distance (0-100%) with 100% equal to a perfect score.
Immediate Post-Concussion Assessment Battery | 8 weeks
  Cognitive assessment-Composite score is generated from each subscale by averaging scores, with 100 being equal to a perfect score.
Driving simulator | 8 weeks
  Reaction time to several scenarios will be measured
Oddball task | 8 weeks
  Number of event related potentials will be measured during responses to stimuli
Flanker task | 8 weeks
  Number of event related potentials will be measured during responses to stimuli
Brain-derived neurotropic factor | 8 weeks
  Saliva will be used to analyze brain-derived neurotropic factor

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Wark, M.D., Principal Investigator — Northern Ontario School of Medicine
Locations (1):
- Fairway Physiotherapy, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT03357042/Prot_SAP_ICF_002.pdf